CLINICAL TRIAL: NCT03105713
Title: Development and Implementation of Surgical Safety Checklists for Patients to Use Before Admission, Before Discharge and After Discharge (PASC) - a Stepped Wedge Cluster Randomized Controlled Trial
Brief Title: Development and Implementation of Patient Safety Checklists Before, During and After In-hospital Surgery
Acronym: PASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Vest (Other); Western Norway University of Applied Sciences (Other); University of Bergen (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: REK Vest (2016/1102)
Record Dates: First submitted 2017-03-20; First posted 2017-04-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Surgery; Safety Issues; Complication; Patient Safety; Health Literacy; Health Economics
Keywords: Checklist; Patient Checklist; Surgery; Safety; Patient Involvement; Undernutrition; Implementation; Health literacy; Health economics
MeSH Terms: conditions — Patient Participation; Malnutrition

STUDY DESIGN:
Intervention Model Description: Stepped Wedge Cluster RCT is considered to align a cross-over design.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All participants are masked for the study outcomes. In intervention arm, the participants are not masked for the checklist intervention.
  Care Providers are masked for patients receiving the intervention and for outcomes.
  Outcome assessors are masked for patients receiving the intervention. Investigators are partially masked for the outcomes across clusters in the intervention phase
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Safety Checklist Intervention (Experimental): The intervention to be administered is a patient safety checklist (two parts) for patients to be performed on paper or electronically: a) before admission to hospital, and b) under hospital stay (discharge)
  Interventions: Other: Patient Safety Checklist
- Controls (No Intervention): Patients do not receive the safety checklist intervention. Care as usual.

INTERVENTIONS:
Other: Patient Safety Checklist — The intervention is developed, validated and to be implemented in seven surgical clusters in two hospitals, in a stepped wedge cluster randomized controlled trial of the PASC for patients to use.
  Arms: Patient Safety Checklist Intervention

SUMMARY:
Building on the Norwegian Patient Safety Program's target areas, the Patients' Surgical Checklist (PASC) will empower surgical patients to become more involved in their own safety and contribute to preventive safety measures. A safety checklist for patients to use has been developed and validated for use in surgical patients. In a Stepped Wedge Cluster RCT effects of patients using their own checklists to avoid preventable patient harm are examined. The project will re-use existing health and personal data collected from patient records and patient reported data as outcome measures. A consortium of all relevant stakeholders and users participate: two hospitals with seven surgical clusters, patient representatives, representatives of general practitioners, and interdisciplinary in-hospital professionals. The important project partners are information and communications technology companies (Helse-Vest IKT and CheckWare service delivery), general practitioners, and national and international research partners leading in the field of patient safety, implementation science and health economics.

DETAILED DESCRIPTION:
The PASC consist of measures that enable patients to optimize their own health prior to surgery and for discharge from hospital. The checklist addresses risk areas as pre-operative information and preparations, post-operative information, and post-operative plans and follow-up. Pre-operative risk areas are contact information, medication safety, health status, optimizing health and nutritional status, dental status, comprehend critical information, preparation two weeks before surgery, communication with surgical ward, and discharge planning. Post-operative risk areas are prevention of complications, medication safety, activity restriction, and pain relief.

The checklist has been developed in cooperation with patients, patients' representatives, surgeons, general practitioners, ward doctors, nurses, pharmacists, clinical nutritionists, safety officers, hospital managers, information technology experts and the researchers. The intervention include paper and electronically versions of the checklist. Of eligible surgical wards, seven were randomly selected based on power calculation. All the invited wards agreed to participate. Surgical patients from these wards, in two Norwegian hospitals, will be invited to participate in the trial. Based on data from a validation and feasibility study of PASC, the power analysis suggest to include 38 patients per month (on average), per cluster over 20 months, as the lowest number of participants to detect a 5% (33.3% relative risk reduction). An intra-cluster-correlation at 0.05, and type I and type II error at 0.05 and 0.20, respectively, were assumed.

The outcomes of this study are primarily patient outcomes (morbidity and mortality). The study further assess outcomes on nutritional status (MST form), implementation (acceptability, appropriateness and feasibility survey), health economic (EQ-5D-3L) data, and health literacy (HLQ), from surveys and forms.

Based on power calculation, 350 questionnaires will be distributed in each arm of the trial (baseline and internvention).

Focus group interviews with content analysis will be applied to assess patients and health care personnel's experiences with patients' use of PASC.

ELIGIBILITY:
Inclusion Criteria:

Elective surgery.

* Age over 18 years.
* Able to use Norwegian language.
* Patients must have had surgery 2-4 weeks before inclusion for the focus group interviews.

Exclusion Criteria:

* Must be cognitive able to use the checklist.
* Age under 18 years.
* Non-surgical procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8559 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Number of complications associated with the participants surgery | Up to 30 days
  Total numbers of complications
Number of complications within respiratory system | Up to 30 days
  Number of respiratory complications
Number of complications within cardio-thoracic system | Up to 30 days
  Number of cardio-thoracic complications
Number of infections | Up to 30 days
  Numbers of infections
Number of nervous system complications | Up to 30 days
  Number of nervous system complications
Volume of bleeding associated with operation | Up to 30 days
  Volume of bleedings in mL
Number of embolism associated with the hospital stay | Up to 30 days
  Number of embolies
Number of mechanical implant complications | Up to 30 days
  Number of mechanical implant complications
Number of re-operations | Up to 30 days
  Number of re-operations
Number of re-admissions | Up to 30 days
  Number of re-admissions

SECONDARY OUTCOMES:
Number of deaths associated with surgery | Up to 90 days
  Total numbers of deaths
Rate of patient scores on Health Literacy Questionaire | Up to 3 months post discharge
  Mean scores of HLQ and EQ5D surveys
Rate of patient scores on EQ5D | Up to 3 months
  Mean scores of EQ5D
Rates of Checklist Implementation Survey scores | Up to 3 months post discharge
  Mean scores on checklist implementation survey

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Klausen, MD, Study Director — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Førde Central Hospital, Førde

IPD SHARING:
Plan to Share IPD: No
REKVest has decided that data which are anonymous, where it directly or indirectly is not possible to identify individuals, could be shared with other scientists or scientific journals.

REFERENCES:
- [Background] Harris K, Softeland E, Moi AL, Harthug S, Ravnoy M, Storesund A, Jurmy E, Skeie E, Waehle HV, Sevdalis N, Haugen AS. Feasibility of implementing a surgical patient safety checklist: prospective cross-sectional evaluation. Pilot Feasibility Stud. 2023 Mar 27;9(1):52. doi: 10.1186/s40814-023-01277-3. PMID 36973815
- [Result] Harris K, Softeland E, Moi AL, Harthug S, Storesund A, Jesuthasan S, Sevdalis N, Haugen AS. Patients' and healthcare workers' recommendations for a surgical patient safety checklist - a qualitative study. BMC Health Serv Res. 2020 Jan 16;20(1):43. doi: 10.1186/s12913-020-4888-1. PMID 31948462
- [Result] Tangvik RJ, Skeie E, Haugen AS, Harthug S, Harris K. Is self-screening for 'at risk of malnutrition' feasible in a home setting? PLoS One. 2024 Apr 16;19(4):e0299305. doi: 10.1371/journal.pone.0299305. eCollection 2024. PMID 38625912
- [Derived] Harris K, Waehle HV, Storesund A, Harthug S, Tangvik RJ, Monsen Lukcova D, Havik W, Humberset A, Stavang E, Hagerup K, Teigland Tepstad A, Sandsbakk Austarheim AK, Healey A, Sevdalis N, Haugen AS. Surgical patients' experiences with the Patients' Safety Checklist (PASC): a qualitative interview study. BMJ Open. 2025 Oct 5;15(10):e105554. doi: 10.1136/bmjopen-2025-105554. PMID 41047253
- See also: The Research Council of Norway's Project Bank description of the PASC project — https://prosjektbanken.forskningsradet.no/en/project/FORISS/320475?Kilde=FORISS&distribution=Ar&chart=bar&calcType=funding&Sprak=no&sortBy=date&sortOrder=desc&resultCount=30&offset=0&Organisasjon.3=HUSEBY+G%C3%85RD+Amund+Huseby
- Available data/document: Study Protocol: 2016/1102 — https://prosjektbanken.forskningsradet.no/en/project/FORISS/320475 — Study protocol version 2.1 is up-loaded in ClinicalTrials.gov along with the SAP. English version of the trial and other relevant information on this study can be accessed by e-mail to arvid.steinar.haugen@helse-bergen.no

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT03105713/SAP_000.pdf